CLINICAL TRIAL: NCT06929611
Title: Comparative Study of the Effect of Continuous Caudal Epidural With General Anaesthesia Versus General Anaesthesia on Intra Operative and Post Operative Analgesic Requirements for Lumbar Fixation
Brief Title: Analgesic Requirements for Lumbar Fixation With General Anaesthesia Versus Continuous Caudal Epidural
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Esraa Abdellatif, Assistant lecturer of anesthesia, intensive care unit and pain management, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Continuous caudal epidural
Record Dates: First submitted 2024-01-29; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Anesthesia, General

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated by computer generated randomization into two equal groups A and B.
  * Group A: Patients doing lumbar fixation with combined continuous caudal epidural and general anaesthesia.
  * Group B: Patients doing lumbar fixation under general anaesthesia (opioid analgesia).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combined continuous caudal epidural and general anaesthesia (Active Comparator): -Patients will be located in the prone position for caudal epidural block.Fluoroscopy will be utilized and a lateral view will be obtained to demonstrate the anatomic boundaries of the sacral canal. A 17- or 18-gauge Tuohy-type needle will be inserted in the midline into the caudal canal. An initial dose of 20 ml of 0.25% bupivacaine will be injected in the caudal canal in order to perform sensory block and spare motor power. Then a dose of 10 ml 0.25% bupivacaine will be injected through the epidural catheter every 1-hour intra operatively and at 0-hour and 1-hour post operative. Then the catheter will be removed 1 hour post operative.
  Interventions: Other: Combined continous caudal epidural with general anaesthesia
- General anaesthesia (opioid analgesia) (Active Comparator): -General anaesthesia will be induced with administration of extra doses of fentanyl as needed according to hemodynamic changes suggesting pain sensation
  Interventions: Other: Combined continous caudal epidural with general anaesthesia

INTERVENTIONS:
Other: Combined continous caudal epidural with general anaesthesia — A 17- or 18-gauge Tuohy-type needle will be inserted in the midline into the caudal canal. An initial dose of 20 ml of 0.25% bupivacaine will be injected in the caudal canal in order to perform sensory block and spare motor power. Then a dose of 10 ml 0.25% bupivacaine will be injected through the epidural catheter every 1-hour intra operatively and at 0-hour and 1-hour post operative then the catheter will be removed 1 hour post operative.
  -The following factors will be assessed:
  1. Intra operative heart rate and blood pressure.
  2. Post operative pain assessment according to numeric pain scale score.
  3. Time to rescue analgesia (intravenous analgesia administered after surgery).Patients with numeric pain scale score ≥ 3 at any point of time, will receive intravenous morphine 5mg.
  4. Estimated blood loss and surgeon satisfaction of surgical field.
  5. Total intra operative and post operative analgesia.
  6. Common complications.

SUMMARY:
In this clinical study, the investigators will justify the current practice of combined continuous caudal epidural with general anaesthesia in adult patients undergoing lumbar fixation versus general anaesthesia. Furthermore, the investigators will determine the analgesic requirement, rescue analgesia, hemodynamic changes and possible complications with continuous caudal epidural analgesia.

DETAILED DESCRIPTION:
* The clinical trial will justify the current practice of combined continuous caudal epidural with general anaesthesia in adult patients undergoing lumbar fixation versus general anaesthesia and using this clinical trial to prove the good analgesic effect of continous caudal epidural and its use to decrease opioid use intra and post operative.
* This clinical trial can trace intra and post operative hemodynamic changes while using continuous caudal epidural.
* This clinical trail will record the possible complications and their incidence of continuous caudal epidural.
* Sample size justification: the expected mean intra-operative narcotic consumption among study groups is 186.5 ± 21.6 µg and 106 ± 16.4 µg.

Sample size of 30 patients per group can detect the difference between two groups with power >90% and alpha error 0.05.

* Statistical analysis: this clinical trial will be carried out using the statistical software program. Description of quantitative data as mean and standard deviation and qualitative data as number and percentage.Comparison between the two groups will be done by using the Chi-square test, independent t-test or Mann-Whitney U-test according to the distribution of data. A p-value less than 0.05 will be considered statistically significant.
* Study Procedures:

Patients will be randomly allocated into two equal groups.

Preoperative setting:

* Pre-operative assessment will be done by accurate history taking, full physical examination, laboratory and radiological investigations. including complete blood count (CBC), liver function test (LFT), kidney function test (KFT), prothrombin time (PT) and partial thromboplastin time (PTT) will be checked.
* All patient will be fasting for 8 hours pre operative.
* All patients will be informed about the study design, objectives and techniques.
* Informed consent will be signed by every patient prior to inclusion in the study.
* All patients will be educated about numeric pain scale score which 0 means no pain and 10 means worst imaginable pain.

Intraoperative setting:

* Standard perioperative monitoring will include pulse oximetry, electrocardiogram, end-tidal carbon dioxide measurement, inhaled volatile agent concentration and non-invasive blood pressure measurement.
* Baseline parameters such as oxygen saturation, systolic, diastolic and mean blood pressure, heart rate will be observed.
* Intravenous line will be inserted.
* For all patients, general anaesthesia will be induced by intravenous route using midazolam 0.04 mg/kg, fentanyl 1 µg/kg, propofol 2 mg/kg, atracurium 0.5 mg/kg.
* This will be followed by endotracheal intubation and mechanical ventilation. Maintenance of anaesthesia will be achieved by isoflurane 1.5% in oxygen and air (50:50) and atracurium 0.1 mg/kg every 20 minutes, so as to maintain end tidal carbon dioxide between 35 to 40 mm Hg.
* Intra operative heart rate and mean blood pressure will be recorded. Estimated blood loss will be determined.

Group A: (continuous caudal epidural with general anaesthesia "study group")

* After induction of anaesthesia as mentioned above, patients will be located in the prone position for caudal epidural block. Sterile skin preparation and draping of the entire region will be completed in the standard fashion.
* Fluoroscopy will be utilized and a lateral view will be obtained to demonstrate the anatomic boundaries of the sacral canal. With fluoroscopy, the caudal canal will appear as a translucent layer posterior to the sacral segments. The median sacral crest will be visualized as an opaque line posterior to the caudal canal. The sacral hiatus will be visualized as a translucent opening at the base of the caudal canal. The coccyx will be seen articulating with the inferior surface of the sacrum. A 17- or 18-gauge Tuohy-type needle will be inserted in the midline into the caudal canal. A feeling of a slight "snap" may be appreciated when the advancing needle pierces the sacrococcygeal ligament. Once the needle reaches the ventral wall of the sacral canal, it will be withdrawn and reoriented, directing it more cranially (by depressing the hub and advancing) for further insertion into the canal. The anteroposterior view will be used once the epidural needle is safely situated within the canal and the epidural catheter will be advanced cephalad. In this projection, the intermediate sacral crests will appear as opaque vertical lines on either side of the midline. The sacral foramina will be visualized as translucent and nearly circular areas lateral to the intermediate sacral crests. Once the correct placement of the needle will be confirmed, a catheter will be inserted into the desired location while depth and position will be confirmed fluoroscopically.
* Before the local anaesthetic will be injected, careful aspiration or passive drainage is essential to exclude an unintentional intravascular or intrathecal needle location. An initial dose of 20 ml of 0.25% bupivacaine will be injected in the caudal canal in order to perform sensory block and spare motor power. Then a dose of 10 ml 0.25% bupivacaine will be injected through the epidural catheter every 1-hour intra operatively and at 0-hour and 1-hour post operative. Then the catheter will be removed 1 hour post operative.

Group B: (general anaesthesia "control group")

-General anaesthesia will be induced as described above with administration of extra doses of fentanyl as needed according to hemodynamic changes suggesting pain sensation.

Post-operative setting:

* After completion of surgery, the residual neuromuscular block will be reversed with injection of neostigmine 0.05 mg/kg and atropine 0.01 mg/kg. When patients become suitable for extubation, with stable hemodynamic and adequate muscle power, thorough oral and endotracheal suction followed by extubation will be done.
* Patients will be nursed in post anaesthesia care unit for monitoring of post operative vital signs and for post operative pain assessment by numeric pain scale score at 0-hour and management accordingly.
* Patients postoperative pain will be followed up at the ward at time interval 0, 1, 2, 4, 6 hours.
* Patients will undergo close monitoring for the first 6 hours after caudal injection for overdose or adverse reactions.
* The following factors will be assessed:

  1. Intra operative heart rate and blood pressure.
  2. Post operative pain assessment according to numeric pain scale score 1-10 as (0= no pain, 10 =worst imaginable pain) and hemodynamic parameters at 0, 1, 2, 4, 6 hours.
  3. Time to rescue analgesia (intravenous analgesia administered after surgery) when the numeric pain scale score is 3 or higher. Patients with numeric pain scale score ≥ 3 at any point of time, will receive intravenous morphine 5mg.
  4. Estimated blood loss and surgeon satisfaction of surgical field.
  5. Total intra operative and post operative analgesia in both groups.
  6. Common complications of caudal block in the postoperative period which include hypotension, bradycardia, lower limb numbness and urinary retention. These complications will be recorded and managed accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Age group: Adult patients from age of 21 years to 60 years
* Sex: Both sexes.
* American Society Association Classification (ASA): patients with ASA classification I, II.
* Elective lumbar fixation surgeries.

Exclusion Criteria:

* Patients refuse to give informed consent.
* Patients younger than 21 or older than 60.
* History of bupivacaine allergy.
* Emergency surgeries.
* Patients who underwent previous spine surgeries of any cause.
* Infection at the site of injection.
* Coagulopathy (acquired, induced, genetic).
* ASA Classification: ASA III, IV.
* Severe aortic stenosis, severe mitral stenosis, hypertrophic obstructive cardiomyopathy.
* Severe hypovolemia, Severe uncorrected anemia.
* Increased intra-cranial pressure (i.e., brain tumor or recent head injury).

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Determining the total amount of fentanyl that will be consumed as intra operative analgesia | during intraoperative period (from induction of anesthesia until recovery from general anaesthesia)
  the amount of fentanyl on micrograms used intra operative for both groups

SECONDARY OUTCOMES:
Determining the total amount of morphine that will be given as analgesia | the first 6 hours post operative
  amount of morphine in mg
Analyzing the numeric pain scale score | the first 6 hours post operative
  Post operative pain assessment according to numeric pain scale score 1-10 as (0= no pain, 10 =worst imaginable pain)
Detecting effect of continuous caudal epidural analgesia on intra operative and post operative on vital data (using heart rate) | intra operative and the first 6 hours post operative
  by detecting heart rate(beat/min.)
Identifying the time to the first demand for rescue analgesia | any time during the first 6 hours post operative
  the time of first dose of morphine post operative

CONTACTS AND LOCATIONS:
Overall Officials: Omar Zafer, MD, Study Director — Faculty of Medicine Ain Shams University; Paula Samaan, MD, Study Director — Faculty of Medicine Ain Shams University; Ahmed El-Hennawy, MD, Study Director — Faculty of Medicine Ain Shams University; Mahmoud Ghallab, MD, Study Director — Faculty of Medicine Ain Shams University
Locations (1):
- Faculty of Medicine , Ain Shams University, Cairo, Abbassia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all data that underlie results in a publication
Supporting Information: Study Protocol, ICF
Time Frame: the data will be available at the end of the study nearly in six months It will be available once the paper of the study is published in a journal
Access Criteria: the data will be shared with any researcher interested in subject

REFERENCES:
- [Background] Hurley WR. Acute postoperative pain.In: Miller RD, Eriksson LI, Fleisher LA, Wiener-Kronish JP, Young WL, editors. Miller's Anesthesia. 7th ed. Philadelphia: Churchill Livingstone. 2010; 2757-81.
- [Background] Kao SC, Lin CS. Caudal Epidural Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:9217145. doi: 10.1155/2017/9217145. Epub 2017 Feb 26. PMID 28337460
- [Background] Schug SA, Bruce J. Risk stratification for the development of chronic postsurgical pain. Pain Rep. 2017 Oct 31;2(6):e627. doi: 10.1097/PR9.0000000000000627. eCollection 2017 Nov. PMID 29392241
- [Background] Waurick K, Waurick R. [History and Technique of Epidural Anaesthesia]. Anasthesiol Intensivmed Notfallmed Schmerzther. 2015 Jul;50(7-8):476-82; quiz 483. doi: 10.1055/s-0041-100845. Epub 2015 Jul 31. German. PMID 26230893
- [Background] Wiegele M, Marhofer P, Lonnqvist PA. Caudal epidural blocks in paediatric patients: a review and practical considerations. Br J Anaesth. 2019 Apr;122(4):509-517. doi: 10.1016/j.bja.2018.11.030. Epub 2019 Feb 1. PMID 30857607
- [Result] Abdel Hady Sarah Mahmoud Farid Mahmoud, Ahmed Azza Youssef Ibrahim, Neamat-Allah Hatem Saaed Abdel Hamid, et al. Combined caudal epidural with general anesthesia for lumbar discectomy. Ain Shams medical journal. 2022; 73(3): 695-704.
- [Result] Al Oweidi AS, Klasen J, Al-Mustafa MM, Abu-Halaweh SA, Al-Zaben KR, Massad IM, Qudaisat IY. The impact of long-lasting preemptive epidural analgesia before total hip replacement on the hormonal stress response. A prospective, randomized, double-blind study. Middle East J Anaesthesiol. 2010 Jun;20(5):679-84. PMID 20803856
- [Result] Barham G, Hilton A. Caudal epidurals: the accuracy of blind needle placement and the value of a confirmatory epidurogram. Eur Spine J. 2010 Sep;19(9):1479-83. doi: 10.1007/s00586-010-1469-8. Epub 2010 May 29. PMID 20512512
- [Result] Benyahia NM, Verster A, Saldien V, Breebaart M, Sermeus L, Vercauteren M. Regional anaesthesia and postoperative analgesia techniques for spine surgery - a review. Rom J Anaesth Intensive Care. 2015 Apr;22(1):25-33. PMID 28913452
- [Result] El-Feky EM and Abd El Aziz AA. Fentanyl, dexmedetomidine, dexamethasone as adjuvant to local anesthetics in caudal analgesia in pediatrics. Egypt J Anaesth. 2015; 31:175-80.
- [Result] Ni Eochagain A, Singleton BN, Moorthy A, Buggy DJ. Regional and neuraxial anaesthesia techniques for spinal surgery: a scoping review. Br J Anaesth. 2022 Oct;129(4):598-611. doi: 10.1016/j.bja.2022.05.028. Epub 2022 Jul 9. PMID 35817613
- [Result] Fawzi HM, Almarakbi WA. Effect of a preemptive caudal dexmedetomidine-bupivacaine mixture in adult patients undergoing a single-level lumbar laminectomy. Ain Shams J Anesthesiol. 2012; 5:223-8.
- [Result] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233
- [Result] Kumar S, Palaniappan JM, Kishan A. Preemptive Caudal Ropivacaine: An Effective Analgesic during Degenerative Lumbar Spine Surgery. Asian Spine J. 2017 Feb;11(1):113-119. doi: 10.4184/asj.2017.11.1.113. Epub 2017 Feb 17. PMID 28243379
- [Result] Lakshminarasimhaiah G, Madabhushi R, Pai KR. Comparison of Epidural Anaesthesia and General Anaesthesia with Caudal Epidural Analgesia for Minimally Invasive Lumbosacral Spine Surgeries. Int J Anesth Pain Med. 2018; 4 :1-3.
- [Result] Nagappa S, Kalappa S, Sridhara RB. Clonidine as an Adjuvant to Caudal Epidural Ropivacaine for Lumbosacral Spine Surgeries. Anesth Essays Res. 2018 Jan-Mar;12(1):240-245. doi: 10.4103/aer.AER_215_17. PMID 29628589

DOCUMENTS (2):
  • Study Protocol (2025-04-09): https://cdn.clinicaltrials.gov/large-docs/11/NCT06929611/Prot_000.pdf
  • Informed Consent Form (2025-04-09): https://cdn.clinicaltrials.gov/large-docs/11/NCT06929611/ICF_001.pdf